CLINICAL TRIAL: NCT02616250
Title: Efficacy and Safety of Ivermectin 1% Topical Cream Associated With Brimonidine 0.33% Topical Gel in the Treatment of Moderate to Severe Rosacea
Brief Title: MirvasO Soolantra Association In the Treatment of Moderate to Severe rosaCea.
Acronym: MOSAIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.03.SPR.105069
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2018-02

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Brimonidine Tartrate; Gels; Ivermectin; Intravital Microscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brimonidine 0.33% gel / CD07805/47 (Br) + Ivermectin 1% cream (Experimental): Half group will receive once-daily Br 0.33% gel in the morning and once-daily IVM 1% cream in the evening for 12 weeks.
  Half group will receive once-daily Br vehicle gel in the morning for the first 4 weeks and once-daily Br 0.33% gel in the morning for the following 8 weeks and once-daily IVM 1% cream in the evening for 12 weeks.
  Interventions: Drug: Brimonidine 0.33% gel (Br); Other: CD07805/47 (Br) placebo gel; Drug: Ivermectin 1% cream (IVM)
- CD07805/47 (Br) placebo gel + CD5024 (IVM) placebo cream (Placebo Comparator): Subjects will receive once-daily Br vehicle gel in the morning and once-daily IVM vehicle cream in the evening for 12 weeks.
  Interventions: Other: CD07805/47 (Br) placebo gel; Other: CD5024 (IVM) placebo cream

INTERVENTIONS:
Drug: Brimonidine 0.33% gel (Br)
  Arms: Brimonidine 0.33% gel / CD07805/47 (Br) + Ivermectin 1% cream
Other: CD07805/47 (Br) placebo gel
Drug: Ivermectin 1% cream (IVM)
  Arms: Brimonidine 0.33% gel / CD07805/47 (Br) + Ivermectin 1% cream
Other: CD5024 (IVM) placebo cream
  Arms: CD07805/47 (Br) placebo gel + CD5024 (IVM) placebo cream

SUMMARY:
The main objective of this study is to evaluate the efficacy of Ivermectin 1% cream (IVM) associated with Brimonidine 0.33% gel (Br) compared with the association of their respective vehicles in the treatment of moderate to severe rosacea.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female subjects age 18 years or older;
2. Subjects with a minimum of 15 but not more than 70 inflammatory lesions (papules and pustules) of rosacea on the face;
3. Subjects with moderate or severe diffuse persistent facial erythema of rosacea (scored 3 or 4 according to Clinician's Erythema Assessment [CEA]);
4. Subjects with moderate or severe papulopustular rosacea (scored 3 or 4 according to the Investigator's Global Assessment [IGA]);
5. Female subjects of childbearing potential with a negative urine pregnancy test (UPT);
6. Female subjects of childbearing potential must practice a highly effective method of contraception during the study;
7. Females subjects of non-childbearing potential;

Main Exclusion Criteria:

1. Subjects with particular forms of rosacea or other concomitant facial dermatoses that may be confounded with rosacea;
2. Subjects with more than 2 nodules of rosacea on the face;
3. Subjects with any uncontrolled chronic or serious disease or medical condition that may either interfere with the interpretation of the clinical trial results, or with optimal participation in the study or would present a significant risk to the subject;
4. Subjects with known or suspected allergies or sensitivities to any component of the investigational and non-investigational products, including the active ingredients brimonidine or salts of brimonidine like brimonidine tartrate and ivermectin;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - Fort Smith, Arkansas
  - Rogers, Arkansas
  - Sacramento, California
  - Orlando, Florida
  - Omaha, Nebraska
  - New York, New York
  - Pflugerville, Texas
- Canada (6):
  - Surrey, British Columbia
  - Markham, Ontario
  - Peterborough, Ontario
  - Richmond Hill, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Brimonidine 0.33% Gel / CD07805/47 (Br) + Ivermectin 1% Cream: Half group will receive once-daily Br 0.33% gel in the morning and once-daily IVM 1% cream in the evening for 12 weeks.
  Half group will receive once-daily Br vehicle gel in the morning for the first 4 weeks and once-daily Br 0.33% gel in the morning for the following 8 weeks and once-daily IVM 1% cream in the evening for 12 weeks.
  Brimonidine 0.33% gel (Br)
  CD07805/47 (Br) placebo gel
  Ivermectin 1% cream (IVM)
- CD07805/47 (Br) Placebo Gel + CD5024 (IVM) Placebo Cream: Subjects will receive once-daily Br vehicle gel in the morning and once-daily IVM vehicle cream in the evening for 12 weeks.
  CD07805/47 (Br) placebo gel
  CD5024 (IVM) placebo cream
Period: Overall Study
Arm/Group | Brimonidine 0.33% Gel / CD07805/47 (Br) + Ivermectin 1% Cream | CD07805/47 (Br) Placebo Gel + CD5024 (IVM) Placebo Cream
Started | 95 | 95
Completed | 85 | 86
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimonidine 0.33% Gel / CD07805/47 (Br) + Ivermectin 1% Cream | CD07805/47 (Br) Placebo Gel + CD5024 (IVM) Placebo Cream | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (14.8) | 48.0 (13.6) | 50.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 67 | 70 | 137

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Variable: Percentage of Patients Defined as Success on the Global Rosacea Severity Grading Scale Called Investigator's Global Assessment (IGA):
Description: Percentage of patients defined as success as per scores of IGA; ie: clear (score=0) or almost clear (score=1)
Time Frame: week 12/Hour 3
Population: Intent To Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Brimonidine 0.33% Gel / CD07805/47 (Br) + Ivermectin 1% Cream | CD07805/47 (Br) Placebo Gel + CD5024 (IVM) Placebo Cream
Number analyzed (Participants) | 95 | 95
Participants | 53 | 35

ADVERSE EVENTS:
Time Frame: All AEs occurring after subject's consent and during the study were recorded; 3 months for a given subject 10 months for the study; ie: from first subject enrolled until last visit of last subject enrolled
Arm/Group | Brimonidine 0.33% Gel / CD07805/47 (Br) + Ivermectin 1% Cream | CD07805/47 (Br) Placebo Gel + CD5024 (IVM) Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/95
Serious Adverse Events (participants affected / at risk) | 5/95 | 1/95
Other Adverse Events (participants affected / at risk) | 8/95 | 13/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brimonidine 0.33% Gel / CD07805/47 (Br) + Ivermectin 1% Cream (N=95) | CD07805/47 (Br) Placebo Gel + CD5024 (IVM) Placebo Cream (N=95)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine 0.33% Gel / CD07805/47 (Br) + Ivermectin 1% Cream (N=95) | CD07805/47 (Br) Placebo Gel + CD5024 (IVM) Placebo Cream (N=95)
Upper respiratory tract infection (Infections and infestations) | 2 | 5
nasopharyngitis (Infections and infestations) | 3 | 5
erythema (Skin and subcutaneous tissue disorders) | 3 | 1
rosacea (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No